CLINICAL TRIAL: NCT02043145
Title: Safety and Efficacy of BOTOX® (Botulinum Toxin Type A) in Korea
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: EPI-MULT-100
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-05

CONDITIONS: Hyperhidrosis; Muscle Spasticity; Glabellar Lines
MeSH Terms: conditions — Hyperhidrosis; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Axillary Hyperhidrosis: Patients with Axillary Hyperhidrosis who are treated with BOTOX® (botulinum toxin Type A) as prescribed according to standard of care in clinical practice.
  Interventions: Biological: botulinum toxin Type A
- Focal Spasticity: Patients with Focal Spasticity who are treated with BOTOX® (botulinum toxin Type A) as prescribed according to standard of care in clinical practice.
  Interventions: Biological: botulinum toxin Type A
- Glabellar Lines: Patients with moderate or severe Glabellar Lines who are treated with BOTOX® (botulinum toxin Type A) as prescribed according to standard of care in clinical practice.
  Interventions: Biological: botulinum toxin Type A

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A (BOTOX®) as prescribed according to standard of care in clinical practice.

SUMMARY:
This post marketing surveillance study in Korea will evaluate the safety and efficacy of BOTOX (botulinum toxin Type A) in patients who receive treatment according to standard of care for primary axillary hyperhidrosis, focal spasticity or moderate to severe glabellar lines in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with BOTOX® (botulinum toxin Type A) as prescribed according to standard of care in clinical practice for primary axillary hyperhidrosis, focal spasticity or moderate to severe glabellar lines.

Exclusion Criteria:

* None.

Ages: 18 Years to 65 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with BOTOX® (botulinum toxin Type A) as prescribed according to standard of care in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 727 (Actual)
Dates: Start 2008-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axillary Hyperhidrosis | Focal Spasticity | Glabellar Lines
Started | 55 | 247 | 425
Completed | 55 | 247 | 425
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline measures were based on the Safety population that included all participants treated with BOTOX® as prescribed. Participants previously treated with survey drug (BOTOX®) were excluded.
Groups:
- Total: Total of all reporting groups
Arm/Group | Axillary Hyperhidrosis | Focal Spasticity | Glabellar Lines | Total
Number analyzed (Participants) | 55 | 237 | 423 | 715
Age, Customized [Number; unit: Participants]
  < 30 years | 24 | 30 | 67 | 121
  30 to 39 years | 21 | 21 | 154 | 196
  40 to 49 years | 6 | 56 | 112 | 174
  >=50 years | 4 | 130 | 90 | 224
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 78 | 376 | 502
  Male | 7 | 159 | 47 | 213

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events (AEs) and Serious Adverse Drug Reactions (SADRs)
Description: An AE was defined as any undesirable changes in medical findings (including laboratory test findings) identified during medical examinations as well as AEs associated with the study drug application that occurred during or after administration of the study drug, regardless of causal relationship to the study drug. A SADR was any drug reaction that: resulted in death or was life threatening, required hospitalization or prolonged hospitalization, caused persistent or significant disability/incapacity, caused a congenital anomaly/birth defect or other medically important event.
Time Frame: 4 Years
Population: Safety population included all participants treated with BOTOX® as prescribed. Participants previously treated with survey drug (BOTOX®) were excluded.
Measure: Number; unit: participants
Arm/Group | Axillary Hyperhidrosis | Focal Spasticity | Glabellar Lines
Number analyzed (Participants) | 55 | 237 | 423
participants
  Adverse Events | 0 | 6 | 5
  Serious Adverse Drug Reactions | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in the Hyperhidrosis Disease Severity Scale (HDSS) Using a 4-Point Scale
Description: Participants assessed their underarm sweat using the 4-point HDSS where: 1=Never noticeable and never interferes with my daily activities, 2=Tolerable but sometimes interferes with my daily activities, 3=Barely tolerable and frequently interferes with my daily activities or 4=Intolerable and always interferes with my daily activities. A negative change from Baseline indicated improvement.
Time Frame: Pre-dose (Baseline), Post-dose (Up to 4 Years)
Population: Efficacy population included all participants who were treated with BOTOX® as prescribed. Participants previously treated with survey drug (BOTOX®), who violated dose/administration or who were missing data were excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Axillary Hyperhidrosis
Number analyzed (Participants) | 54
score on a scale
  Pre-dose (Baseline) | 2.93 (0.72)
  Change from Baseline at Post-dose | -1.61 (0.79)

3. Primary Outcome: Change From Baseline in the Modified Ashworth Scale (MAS) Using a 6-Point Scale
Description: The MAS assessed the degree of muscle tone during movement of the upper limbs compared to normal muscle tone using a 6-point scale at where: 0=no increase in muscle tone, 1=Slight increase in muscle tone manifested by a catch and release or by minimal resistance at the end of the range of motion when the part is moved, 1+=Slight increase in muscle tone manifested by a catch followed by minimal resistance throughout the remainder of the range of motion, 2=Marked increase in muscle tone through most of the range of motion but affected part easily moved, 3=Considerable increase in muscle tone passive movement difficult or 4=Affected part rigid in movement or extension. A low score indicated little or no stiffness (best). A high score indicated severe stiffness (worse). A negative change from Baseline indicated improvement.
Time Frame: Pre-dose (Baseline), Post-dose (Up to 4 Years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Focal Spasticity
Number analyzed (Participants) | 167
score on a scale
  Pre-dose (Baseline) | 2.85 (0.73)
  Change from Baseline at Post-dose | -1.22 (0.64)

4. Primary Outcome: Change From Baseline in the Investigator Assessment of Glabellar Line Severity Using a 4-point Scale
Description: The Investigator assessed the severity of the patient's glabellar lines at maximum frown using the 4-point Facial Wrinkle Scale (FWS) where: 0=none, 1=mild, 2=moderate or 3=severe. A negative change from Baseline indicated improvement.
Time Frame: Pre-dose (Baseline), Post-dose (Up to 4 Years)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Glabellar Lines
Number analyzed (Participants) | 383
score on a scale
  Pre-dose (Baseline) | 2.27 (0.56)
  Change from Baseline at Post-dose | -1.53 (0.54)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected for Up to 4 Years
Description: Safety population, all participants treated with BOTOX® as prescribed excluding participants previously treated with survey drug (BOTOX®), was used to assess the number of participants at risk for Adverse Events and Serious Adverse Events.
Arm/Group | Axillary Hyperhidrosis | Focal Spasticity | Glabellar Lines
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/237 | 0/423
Other Adverse Events (participants affected / at risk) | 0/55 | 0/237 | 0/423

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.